CLINICAL TRIAL: NCT03118219
Title: Positive Adjustment in Case of Involuntary Childlessness - a Smartphone-supported Intervention Study as RCT
Brief Title: Positive Adjustment Coping Intervention
Acronym: PACI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Maren Schick, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-074/2017
Record Dates: First submitted 2017-03-29; First posted 2017-04-18 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Infertility/Sterility
Keywords: assisted reproductive technology; embryo transfer; online intervention; rct
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive adjustment coping intervention (Experimental): All persons allocated to the intervention group will receive daily text messages (SMS) to their smartphones with sentences for positive adjustment over two weeks starting from the day of the egg-cell punctuation.
  Interventions: Other: Positive adjustment coping intervention
- Brainteaser (Other): All persons allocated to the comparison intervention group will receive daily text messages (SMS) to their smartphones with brainteasers over two weeks starting from the day of the egg-cell punctuation.
  Interventions: Other: Brainteaser

INTERVENTIONS:
Other: Positive adjustment coping intervention — see arm description
  Arms: Positive adjustment coping intervention
Other: Brainteaser — see arm description
  Other Names: Comparison intervention group
  Arms: Brainteaser

SUMMARY:
Involuntary childlessness is experienced as emotionally stressful, however psychosocial counseling is not always available on the spot. Aim of this RCT study is to examine the efficacy and acceptance of a psychological low-dose online intervention for couples in reproductive treatment.

DETAILED DESCRIPTION:
About 8% of all couples of reproductive age are involuntary childless, and just about 25,000 couples receive a medical treatment each year in Germany, which is experienced as "roller coaster of emotions". The positive effect of "face-to-face" counseling for couples with a desire for children has been proven. However, this does not yet apply to a variety of other forms of intervention, e.g. telephone or online counseling.

In this study, the effectiveness of a smartphone-supported psychosocial intervention for women and men in reproductive treatment will be examined in a randomized controlled pre-post design.

For this purpose, an intervention group and a comparison intervention group of each n = 60 couples in reproductive treatment will be examined at two points during a four-week interval using the ScreenIVF questionaire. The ScreenIVF will be completed paper-pencil before the intervention and online after the intervention. In the fourteen-day waiting period between oocyte puncture and pregnancy test (or the reappearance of menstruation), both groups receive either positive adjustment techniques or brainteasers.In addition, both groups are questioned one month after the post-measurement date on the perceived effectiveness and practicability of the intervention techniques.

Sociodemographic variables (such as age, education) and medical data (such as diagnosis, previous treatment cycles) as potential moderators, as well as possible pregnancies at the second measurement time will be reported.

No adverse effects or other risks are expected for the study participants.

ELIGIBILITY:
Inclusion Criteria:

All couples undergoing infertility treatment (in vitro fertilization or intracytoplasmic sperm injection) at the Department of Gynecologic Endocrinology and Fertility Disorders at Heidelberg University Women's Hospital, which have

* agreed to participate in the study
* indicated their mobile phone number
* sufficient knowledge of German language.

If one partner is refusing to participate, the other person may be admitted as an individual.

Exclusion Criteria:

* denial of participation
* non-existent smartphone
* insufficient knowledge of German language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Differences in the Screen IVF questionaire between the intervention groups | through study completion, an average of 2 years
  Differences in the ScreenIVF risk profile at post-measurement time between the intervention group of positive adjustment and the intervention comparison group with the brainteasers

SECONDARY OUTCOMES:
Quantitative evaluation of participants' opinion about the intervention | through study completion, an average of 2 years
  Participants will be questioned about the perceived effectiveness and practicability of the intervention techniques with quantitative items (Rating scales).
Qualitative evaluation of participants' opinion about the intervention | through study completion, an average of 2 years
  Participants will be questioned about the recommendations to others concerning the intervention techniques (open questions)

CONTACTS AND LOCATIONS:
Overall Officials: Tewes Wischmann, PD Dr., Study Director — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lancastle D, Boivin J. A feasibility study of a brief coping intervention (PRCI) for the waiting period before a pregnancy test during fertility treatment. Hum Reprod. 2008 Oct;23(10):2299-307. doi: 10.1093/humrep/den257. Epub 2008 Jul 15. PMID 18628259
- [Derived] Kremer F, Schick M, Roesner S, Germeyer A, Moessner M, Bauer S, Ditzen B, Wischmann T. Smartphone-supported Positive Adjustment Coping Intervention (PACI) for couples undergoing fertility treatment: A randomised controlled trial. PLoS One. 2025 Dec 8;20(12):e0335776. doi: 10.1371/journal.pone.0335776. eCollection 2025. PMID 41359611
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Schick M, Roesner S, Germeyer A, Moessner M, Bauer S, Ditzen B, Wischmann T. Smartphone-supported Positive Adjustment Coping Intervention (PACI) for couples undergoing fertility treatment: a randomised controlled trial protocol. BMJ Open. 2019 Jul 9;9(7):e025288. doi: 10.1136/bmjopen-2018-025288. PMID 31289056